CLINICAL TRIAL: NCT04922645
Title: A Multicenter, Randomized, Open-label, Active-controlled Study to Assess the Impact of Auryxia (Ferric Citrate) on Erythropoiesis-Stimulating Agent (ESA) Use, Intravenous (IV) Iron Use, Phosphate Control, and Anemia Control in Adult Participants on In-Center Hemodialysis or Home Dialysis
Brief Title: Auryxia (Ferric Citrate) Therapy for In-Center and Home Dialysis Participants
Acronym: IMPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: USRC Kidney Research (Network)
Collaborators: Akebia Therapeutics Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USRC-2021-001
Record Dates: First submitted 2021-06-08; First posted 2021-06-10 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Hyperphosphatemia; Anemia, Iron Deficiency; Renal Insufficiency
MeSH Terms: conditions — Hyperphosphatemia; Anemia, Iron-Deficiency; Renal Insufficiency | interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric citrate (commercially available, Auryxia) (Experimental): Ferric citrate, (commercially available Auryxia), supplied as tablets for oral administration containing 1 gram ferric citrate (210 milligrams of ferric iron). Administered orally with meals or snacks.
  Interventions: Drug: Ferric Citrate 1 gram Oral Tablet
- Standard of care phosphate lowering therapy (Active Comparator): Non-Auryxia phosphate-lowering therapy administered as standard of care.
  Interventions: Drug: Standard of care phosphate-lowering therapy

INTERVENTIONS:
Drug: Ferric Citrate 1 gram Oral Tablet — Ferric citrate is an iron-based phosphate binder for the treatment of hyperphosphatemia in subjects with dialysis-dependent chronic kidney disease (DD CKD) and for the treatment of iron deficiency anemia (IDA) in subjects with non-dialysis dependent chronic kidney disease (NDD CKD).
  Other Names: Auryxia
  Arms: Ferric citrate (commercially available, Auryxia)
Drug: Standard of care phosphate-lowering therapy — Subjects randomized to SOC will continue their currently prescribed dose of phosphate lowering therapy which will be dosed per local standard of care to achieve community target serum phosphate goals.
  Arms: Standard of care phosphate lowering therapy

SUMMARY:
This study is being conducted to demonstrate the effect of Auryxia, when used as the primary phosphate lowering therapy, on the overall cumulative use of erythropoiesis-stimulating agent and intravenous iron as well as on the laboratory parameters indicative of phosphate and anemia management.

DETAILED DESCRIPTION:
Approximately 200 participants will be randomized 1:1 (stratified by modality and hemoglobin level) to receive either Auryxia or standard of care phosphate lowering therapy to determine the impact of Auryxia when used as the primary phosphate lowering therapy as compared to standard of care on the utilization of erythropoiesis-stimulating agent and intravenous iron in both in-center and home dialysis populations. This study will also seek to determine the impact of Auryxia, when used as the primary phosphate lowering therapy versus standard of care, on the biochemical assessments of serum phosphate and hemoglobin in both in-center and home dialysis populations.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants greater or equal to 18 years old.
2. Diagnosis of end-stage kidney disease and receiving maintenance dialysis (in-center, home hemodialysis or peritoneal dialysis) for greater or equal to 12 weeks prior to randomization.
3. Most recent transferrin saturation less than or equal to 50 percent
4. Most recent serum phosphate is greater or equal to 3.0 milligrams per deciliter
5. Receiving treatment for greater or equal to 8 weeks prior to screening with non-Auryxia phosphate lowering therapy. No requirement for stable dosing within this time frame.
6. Receiving treatment for greater or equal to 8 weeks prior to screening with erythropoiesis-stimulating agent (any dose, any type). No requirement for stable dosing within this time frame.
7. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

Exclusion Criteria:

1. A known allergy or intolerance to Auryxia or any of its constituents.
2. Hypersensitivity reaction to previous oral iron therapy.
3. History of hemochromatosis or other iron overload syndrome.
4. Active malignancy requiring current treatment except for non-melanoma skin cancer regardless of treatment.
5. Active drug or alcohol dependence or abuse (excluding tobacco use or medicinal or recreational marijuana) within the 12 months prior to Screening or evidence of such abuse (in the opinion of the Investigator).
6. Limited life expectancy (less than 6 months), (in the opinion of the Investigator).
7. Scheduled organ transplant and participants on the kidney transplant wait-list who are expected to receive a transplant within 6 months of screening. Being active on transplant list is not an exclusion. Previous kidney transplant is not an exclusion.
8. Unable to comply with study requirements or in the opinion of the Investigator not clinically stable to participate in the study.
9. Females who are known to be pregnant or are breast-feeding during Screening or are planning to become pregnant and breastfeeding during the study period.
10. Evidence of clinically active infection at the time of Screening.
11. Use of an investigational medication or participation in an investigational study within 30 days prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Difference in mean dose of erythropoiesis-stimulating agent (standardized Units per month) between Auryxia and standard of care treatment groups | Baseline period (Month -3 to Day 1) to months 4to 6 (efficacy evaluation period)
  Difference in change from baseline period (Month -3 to Day 1) to months 4 to 6 (efficacy evaluation period) in mean dose of erythropoiesis-stimulating agent (standardized Units per month) between Auryxia and standard of care treatment groups.
Difference in mean dose of intravenous iron (milligram per month) between Auryxia and standard of care treatment groups. | Baseline period (Month -3 to Day 1) to months 4 to6 (efficacy evaluation period)
  Difference in change from baseline period to efficacy evaluation period in mean dose of intravenous iron (milligrams per month) between Auryxia and standard of care treatment groups.

SECONDARY OUTCOMES:
Difference in hemoglobin measurements | Baseline period (Month -3 to Day 1) to months 4to6 (efficacy evaluation period).
  Difference in proportion of measurements with hemoglobin at or above 10.0 grams per deciliter between Auryxia and standard of care treatment groups during efficacy evaluation period.
Difference in serum phosphate measurements | Baseline period (Month -3 to Day 1) to months 4to6 (efficacy evaluation period)
  Difference in proportion of measurements with serum phosphate at or below 5.5 milligrams per deciliter between Auryxia and standard of care treatment groups during efficacy evaluation period.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - US Renal Care - Dimond, Anchorage, Alaska
  - US Renal Care - Mesa, Mesa, Arizona
  - US Renal Care - Pine Bluff, Pine Bluff, Arkansas
  - US Renal Care - Northridge Roscoe, Granada Hills, California
  - US Renal Care - Dalton, Dalton, Georgia
  - US Renal Care - Major Health, Shelbyville, Indiana
  - US Renal Care - Red Rocks, Gallup, New Mexico
  - US Renal Care - North Dallas, Dallas, Texas
  - Dallas Renal Group, Dallas, Texas
  - US Renal Care - Houston Street, San Antonio, Texas
  - US Renal Care - Palo Alto, San Antonio, Texas
  - US Renal Care - Pleasanton Rd., San Antonio, Texas
  - US Renal Care - Westover Hills, San Antonio, Texas

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086